CLINICAL TRIAL: NCT05179928
Title: Is Erector Spinae Plane Block More Effective Than Rectus Sheath Block for Postoperative Analgesia After Supraumbilical Surgery in Adult Patients
Brief Title: Erector Spinae Plane Block Versus Rectus Sheath Block for Postoperative Analgesia After Supraumbilical Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DTH: 21004
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Post Operative Pain
Keywords: Erector Spinae Plane Block; Rectus Sheath Block; Regional Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (n=30) (Active Comparator): Erector Spinae Plane Block
  Interventions: Procedure: Erector Spinae Plane Block (ESPB)
- Group R (n=30) (Active Comparator): Rectus Sheath Block
  Interventions: Procedure: Rectus Sheath Block (RSB)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESPB) — Postoperative Bilateral Ultrasound-guided ESPB
  Arms: Group E (n=30)
Procedure: Rectus Sheath Block (RSB) — Postoperative Bilateral Ultrasound-guided RSB
  Arms: Group R (n=30)

SUMMARY:
Objectives: To compare the effectiveness of erector spinae plane block (ESPB) and rectus sheath block (RSB) in providing postoperative analgesia after supraumbilical surgery in adult patients and their impact on the patient's outcomes.

Background: Supraumbilical surgery for hernia repair is the second-most-popular after surgical inguinal hernia repair and is accompanied by moderate to severe postoperative pain, so patients always require large doses of opioids within the first postoperative day. Because opioids have several adverse effects such as drowsiness, pruritus, nausea, and vomiting, regional analgesic techniques are an essential component of postoperative opioid-sparing analgesia. Previous studies have shown that regional analgesic techniques after abdominal wall surgeries can be an essential element of a postoperative pain management strategy with minimal adverse effects and hemodynamic responses.

ESPB provides both somatic and visceral analgesia to the abdominal wall, through the blockade of the anterior rami of spinal nerves and the rami communicants involving sympathetic nerve fibers. RSB provides analgesia to the anterior abdominal wall from the xiphoid process to the symphysis pubis, through the blockade of the anterior rami of the 7th to 12th intercostal nerves. The dermatomal distribution of ESPB and RSB makes them ideal regional analgesic techniques after abdominal surgery, and to our knowledge, there were no previous trials that studied the difference between them.

Patients and Methods: This was a prospective, randomized (1:1), double-blind clinical trial on 60 patients scheduled for elective supraumbilical surgery under general anesthesia at our hospital. Patients will be randomly allocated into two equal groups (30 patients each) and will receive: in group E; general anesthesia with postoperative bilateral ultrasound-guided ESPB, whereas in group R; general anesthesia with postoperative bilateral ultrasound-guided RSB.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 60 years
* Body Mass Index (BMI) < 35 kg/m²

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status > II
* Age < 21 years or > 60 years
* Body Mass Index (BMI) ≥ 35
* Local infection at the puncture site
* Altered mental status
* Pregnant women
* Allergy to study drugs
* Chronic pain
* Coagulation abnormalities or on anticoagulants
* Severe hepatic or kidney disease

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean and Standard deviation of time to the first request of postoperative rescue analgesic (minutes) (mean±SD) | 24 hours after block performance
  The time interval between the block performance and the first request of postoperative analgesia

SECONDARY OUTCOMES:
Mean and Standard deviation of Numeric Pain Rating Scale (NPRS) score (mean±SD) | 24 hours after block performance
  NPRS measures the severity of postoperative pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (30 minutes, 1h, 6h, 12h, 18h, 24h) after block performance
Mean and Standard deviation of the total dose of the rescue analgesic consumed (milligrams) (mean±SD) | 24 hours after block performance
  The total dose of the rescue analgesic consumed in the first 24 hours after block performance
Number of participants and Rate of Postoperative Complications | 24 hours after block performance
  Number of participants and Rate of: Nausea, Vomiting, Hematoma formation, Bowel perforation, and Pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt